CLINICAL TRIAL: NCT05987462
Title: Effects of a 12 Week Green Walking Intervention on Body Mass Index, Lipids Profile, Disease Perception, and Quality of Life in Patients With Myocardial Infarction: A Quasi-Experimental Study
Brief Title: The Effect of Green Walking on Myocardial Infarction Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AYNUR CİN (Other)
Responsible Party: Sponsor-Investigator, AYNUR CİN, ASST. PROF. DR, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KTU-ACIN-9286
Record Dates: First submitted 2023-07-02; First posted 2023-08-14 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction; Quality of Life
Keywords: Disease; Nature; Perception; Quality of Life; Green Walking; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; Disease

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Walk group (Experimental): Patients who were admitted to the Cardiology Outpatient Clinic of Y State Hospital and passed the 6MWT conducted by the cardiology physician were eligible for participation in the green walk group. Following the physician's examination at the Cardiology Outpatient Clinic, the researcher conducted face-to-face interviews with the patients in a private room. During these interviews, the patients were administered the Structured Patient Information Form, Blood Lipids and BMI Monitoring Form, the Brief IPQ, and the MIDAS, and the collected data were recorded on the respective forms. Then, the researcher provided detailed information to the patients about green walking. For the randomized MI patients, two groups were formed, and they engaged in a 50-minute green walking three days a week for 12 weeks, under the guidance of the researcher. The green walk group's walks were scheduled differently for the two subgroups.
  Interventions: Other: Green walking
- Control group (No Intervention): Patients who were admitted to the Cardiology Outpatient Clinic of X State Hospital and passed the 6MWT conducted by the cardiology physician were enrolled in the control group. Upon their visit to the outpatient clinic, the patients in this group underwent a face-to-face interview, during which they were administered the "Structured Patient Information Form," the "Blood Lipids and BMI Monitoring Form," the "Brief-IPQ," and the "MIDAS" as pretests. . The patients in the control group continued with their routine daily activities. No specific intervention or additional measures were implemented by the investigator in this group. Furthermore, a follow-up "Blood Lipids and BMI Monitoring Form" was administered to the patients during their visit to the Cardiology Outpatient Clinic in the middle of the study (6th week). At the end of the 12-week period, the patients in the control group underwent a posttest.

INTERVENTIONS:
Other: Green walking — The researcher provided detailed information to the patients about green walking. For the randomized MI patients, two groups were formed, and they engaged in a 50-minute green walking three days a week for 12 weeks, under the guidance of the researcher. The green walk group's walks were scheduled differently for the two subgroups. The first subgroup had their 50-minute walk on Monday, Wednesday, and Saturday, while the second subgroup had their walks on Tuesday, Thursday, and Sunday. This arrangement ensured a standardized time interval between green walks for both groups.
  Arms: Green Walk group

SUMMARY:
In this quasi-experimental study, which involved having patients who had experienced a MI engage in 50 minute green walks three times a week for 12 weeks, the following hypotheses were tested: High-intensity interval green walking has the effect of reducing the anthropometric measurements of patients undergoing MI. High-intensity interval green walking has the effect of reducing LDL, triglyceride, total cholesterol levels and increasing HDL levels of patients who have with MI. High-intensity interval green walking has a positive effect on the perception of disease of patients who have undergone MI. High-intensity interval green walking has an effect on improving the quality of life of patients with MI.

Research Question 1: What is the impact of green walking on the body mass index (BMI) of patients with MI? Research Question 2: How does green walking influence blood lipid levels (triglycerides, LDL, total cholesterol, and HDL) in patients with MI? Research Question 3: What is the effect of green walking on the perception of the disease in patients with MI? Research Question 4: How does green walking affect the quality of life of patients with MI? 2 Groups: Green walking group and control group

DETAILED DESCRIPTION:
Setting and Time of the Study: The study population consisted of patients who were receiving outpatient care at the Cardiology Outpatient Clinic of X and Y State Hospital and had experienced a MI at least three months ago. To determine the appropriate sample size, a power analysis was conducted using the G*Power 3.1.9.6 program based on a previous study involving MI patients. The power analysis resulted in a sample size of 34 patients in total, with 17 patients allocated to each group. This sample size was determined to achieve 80% power, an effect size of 0.87, and a margin of error of 5%. However, considering that increasing the sample size would decrease the standard error and increase the study power, each group was increased by 75%. As a result, a total of 60 patients, with 30 patients in each group, were included in the study.

Due to the limited availability of myocardial infarction (MI) patients residing near green walking environments suitable for the intervention, participants in the experimental group were selected based on their geographical proximity to such areas. These 30 patients were receiving outpatient care at the Cardiology Outpatient Clinic of Y State Hospital and had experienced an MI at least three months prior. In contrast, the control group consisted of 30 MI patients from X State Hospital, located in an urban setting without access to green walking spaces, also selected based on outpatient follow-up and a history of MI at least three months earlier.Random assignment was not feasible due to logistical constraints related to the participants' residential locations. Instead, criterion sampling was used, whereby individuals meeting predefined inclusion criteria were selected. Although randomization was not possible, considerable efforts were made to ensure the comparability of the two groups. Both hospitals had similar infrastructures, were staffed by specialist cardiologists, and served populations with comparable demographic characteristics. Statistical analyses confirmed no significant differences between groups in terms of demographic and clinical variables, supporting the assumption of group equivalence. Additionally, both groups engaged in high-intensity intermittent physical activity, ensuring similarity in baseline activity levels.

Green Walk Group: The written consents of the green walking group were obtained before starting the study after the doctor's declaration was received. Patients who were admitted to the Cardiology Outpatient Clinic of Y State Hospital and passed the 6MWT conducted by the cardiology physician were eligible for participation in the green walk group. Following the physician's examination at the Cardiology Outpatient Clinic, the researcher conducted face-to-face interviews with the patients in a private room. During these interviews, the patients were administered the Structured Patient Information Form, Blood Lipids and BMI Monitoring Form, the Brief IPQ, and the MIDAS, and the collected data were recorded on the respective forms. Then, the researcher provided detailed information to the patients about green walking. Patients' choice of walking shoes before going on a green walk, whether their shoelaces are tied, whether they are wearing shoes of the appropriate size, etc. checked by the researcher. The researcher had a first aid kit (a patch, bandage, elastic bandage, large triangular bandage, cold compress bag, cotton, band-aid, disposable gloves, scissors, tweezers, pocket knife, vaseline, hand sanitizer, antiseptic solution, surgical mask, waste bag) ready for health problems that may develop during the green walking process. The green walking group was divided into two groups by the block randomization method. For the randomized MI patients, two groups were formed, and they engaged in a 50-minute green walking three days a week for 12 weeks, under the guidance of the researcher. The area close to the district center, easy to reach, passing by a stream and surrounded by trees was determined as a walking path. The walking path was two km long. Patients constantly used the same route for a green walking. A green walking track with a slope-free difficulty rating of one was selected, which is suitable for patients who have had a MI. Small gifts were given to encourage patients' participation in the green walking. The green walk group's walks were scheduled differently for the two subgroups. The first subgroup had their 50-minute walk on Monday, Wednesday, and Saturday, while the second subgroup had their walks on Tuesday, Thursday, and Sunday. This arrangement ensured a standardized time interval between green walks for both groups. Additionally, a follow-up Blood Lipids and BMI Monitoring Form was administered to the patients during their visit to the Cardiology Polyclinic in the middle of the study (6th week). At the end of the 12-week period, the patients in the green walk group underwent a posttest evaluation.

Control Group: The written consents of the control walking group were obtained before starting the study. Patients who were admitted to the Cardiology Outpatient Clinic of X State Hospital and passed the 6MWT conducted by the cardiology physician were enrolled in the control group. Upon their visit to the outpatient clinic, the patients in this group underwent a face-to-face interview, during which they were administered the "Structured Patient Information Form," the "Blood Lipids and BMI Monitoring Form," the "Brief-IPQ," and the "MIDAS" as pretests. The information and data collected from these interviews were recorded on the respective forms. The patients in the control group continued with their routine daily activities. No specific intervention or additional measures were implemented by the investigator in this group. The researcher interacted with the patients in the control group during their Cardiology Polyclinic visits and answered the patients' questions. Furthermore, a follow-up "Blood Lipids and BMI Monitoring Form" was administered to the patients during their visit to the Cardiology Outpatient Clinic in the middle of the study (6th week). At the end of the 12-week period, the patients in the control group underwent a posttest.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being 18 years of age or older,
* being able to communicate verbally,
* being literate,
* having had MI at least three months ago,
* being followed up as an outpatient with the diagnosis of MI in the cardiology outpatient clinic of X state hospital and Y state hospital,
* achieving the six-minute walk test (6MWT),
* having no obstacle to walking (musculoskeletal problems, joint problems, fracture, neuropathy, chronic severe pain, limb loss)
* volunteering to participate in the study.

Exclusion Criteria:

* having blood pressure above 140/90 mmHg or below 90/60 mmHg,
* having active chest pain, dyspnea, bradycardia, or tachycardia, a psychiatric diagnosis, visual, hearing,
* cognitive impairment,
* a balance problem,
* using a walker while walking,
* having Parkinson's disease, dementia, or cancer,
* having undergone any surgery that would prevent walking,
* refusing to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The Structured Patient Information Form | 1 day before the study
  Developed by the researcher after reviewing the literature, the form consisted of two parts. The first part included six questions to determine the sociodemographic characteristics of the patients (gender, age, education level, marital status, employment status, and occupation), and the second part included a total of 10 questions, including four questions to determine the characteristics related to the disease (when MI occurred, presence of MI risk factors, etc.).
The Blood Lipids and BMI Monitoring Form | 1 day before the study
  This form was developed by the researcher in line with the literature. It included blood lipids (HDL, LDL, Triglyceride and Total cholesterol), height (cm), and weight (kg) measurements of the patients. BMI was calculated by dividing body weight by the square meter of height (BMI=kg/m2). The blood lipid measurement results of the patients (1st-week measurement; 6th-week interim measurement; 12th-week measurement) were obtained from the patient file by the researcher during Cardiology Outpatient Clinic visits.
The Brief Illness Perception Questionnaire (Brief IPQ) | 1 day before the study
  This scale was developed by Broadbent et al. in 2006. The nine-item section of the scale defines the emotional and cognitive aspects of illness perception. Each item in the scale consists of open-ended questions and is scored between 0 and 10. In the last item, the individual is asked to indicate three factors that he/she thinks are the cause of his/her illness. These items include consequences, timeline, personal control, treatment control, identity, illness concern, coherency, and emotional response, respectively. The highest and lowest scores are 80 and 0. On the scale, the positive reaction consists of the score given to three sub-dimensions (3rd, 4th, and 7th) with a score between 0-10, and the negative reaction consists of the score given to five sub-dimensions (1st, 2nd, 5th, 6th, and 8th). Sub-dimension (1st, 2nd, 5th, 6th, and 8th) items are reverse scored. High scores indicate a negative perception of illness.
The Myocardial Infarction Dimensional Assessment Scale (MIDAS) | 1 day before the study
  The Turkish validity and reliability of the MIDAS, devised by David Thompson et al. in 2002, were examined by Uysal et al. (2008), and the Cronbach alpha value of the scale was calculated as 0.83. The scale includes 35 items and seven sub-dimensions, including physical activity, insecurity, emotional reaction, dependency, diet, concerns over medication, and side effects. The scoring of the scale is between 0 and 100. A high score on the scale indicates poor health status.
Weight | 1 day before the study
  Weight was measured with a medical scale with a hospital-calibrated height scale while the patients were fasting, after removing their thick clothes and before the physician examination.Then it was recorded The Blood Lipids and BMI Monitoring Form.
Height | 1 day before the study
  Height measurements were performed with the patient standing barefoot with the head in the Frankfort plane and the feet side by side in a medical basin with a height meter calibrated by the hospital.Then it was recorded The Blood Lipids and BMI Monitoring Form.
Body Mass Index | 1 day before the study
  BMI was calculated by dividing body weight by the square meter of height (BMI=kg/m2). Then it was recorded The Blood Lipids and BMI Monitoring Form.
Six-minute walk test | 1 day before the study
  It is a widely used test to assess treatment response in moderately severe heart or lung disease or to assess functional capacity, which is a determinant of mortality and morbidity in a person with a one-time measurement (in diseases such as Alzheimer's, elderly patients, MS, Parkinson's, osteoarthritis, spinal cord injury, stroke).

SECONDARY OUTCOMES:
The Blood Lipids and BMI Monitoring Form | in the middle of the study (6th week).
  This form was developed by the researcher in line with the literature. It included blood lipids (HDL, LDL, Triglyceride and Total cholesterol), height (cm), and weight (kg) measurements of the patients. BMI was calculated by dividing body weight by the square meter of height (BMI=kg/m2). The blood lipid measurement results of the patients (1st-week measurement; 6th-week interim measurement; 12th-week measurement) were obtained from the patient file by the researcher during Cardiology Outpatient Clinic visits.
Weight | in the middle of the study (6th week).Then it was recorded The Blood Lipids and BMI Monitoring Form.
  Weight was measured with a medical scale with a hospital-calibrated height scale while the patients were fasting, after removing their thick clothes and before the physician examination.
Height | in the middle of the study (6th week).
  Height measurements were performed with the patient standing barefoot with the head in the Frankfort plane and the feet side by side in a medical basin with a height meter calibrated by the hospital.Then it was recorded The Blood Lipids and BMI Monitoring Form.
Body Mass Index | in the middle of the study (6th week).
  BMI was calculated by dividing body weight by the square meter of height (BMI=kg/m2). Then it was recorded The Blood Lipids and BMI Monitoring Form.

OTHER OUTCOMES:
The Blood Lipids and BMI Monitoring Form | At the end of the 12-week period
  This form was developed by the researcher in line with the literature. It included blood lipids (HDL, LDL, Triglyceride and Total cholesterol), height (cm), and weight (kg) measurements of the patients. BMI was calculated by dividing body weight by the square meter of height (BMI=kg/m2). The blood lipid measurement results of the patients (1st-week measurement; 6th-week interim measurement; 12th-week measurement) were obtained from the patient file by the researcher during Cardiology Outpatient Clinic visits.
The Brief Illness Perception Questionnaire (Brief IPQ) | At the end of the 12-week period
  This scale was developed by Broadbent et al. in 2006. The nine-item section of the scale defines the emotional and cognitive aspects of illness perception. Each item in the scale consists of open-ended questions and is scored between 0 and 10. In the last item, the individual is asked to indicate three factors that he/she thinks are the cause of his/her illness. These items include consequences, timeline, personal control, treatment control, identity, illness concern, coherency, and emotional response, respectively. The highest and lowest scores are 80 and 0. On the scale, the positive reaction consists of the score given to three sub-dimensions (3rd, 4th, and 7th) with a score between 0-10, and the negative reaction consists of the score given to five sub-dimensions (1st, 2nd, 5th, 6th, and 8th). Sub-dimension (1st, 2nd, 5th, 6th, and 8th) items are reverse scored. High scores indicate a negative perception of illness.
The Myocardial Infarction Dimensional Assessment Scale (MIDAS) | At the end of the 12-week period
  The Turkish validity and reliability of the MIDAS, devised by David Thompson et al. in 2002, were examined by Uysal et al. (2008), and the Cronbach alpha value of the scale was calculated as 0.83. The scale includes 35 items and seven sub-dimensions, including physical activity, insecurity, emotional reaction, dependency, diet, concerns over medication, and side effects. The scoring of the scale is between 0 and 100. A high score on the scale indicates poor health status.
Weight | At the end of the 12-week period
  Weight was measured with a medical scale with a hospital-calibrated height scale while the patients were fasting, after removing their thick clothes and before the physician examination.Then it was recorded The Blood Lipids and BMI Monitoring Form.
Height | At the end of the 12-week period
  Height measurements were performed with the patient standing barefoot with the head in the Frankfort plane and the feet side by side in a medical basin with a height meter calibrated by the hospital.Then it was recorded The Blood Lipids and BMI Monitoring Form.
Body Mass Index | At the end of the 12-week period
  MI was calculated by dividing body weight by the square meter of height (BMI=kg/m2). Then it was recorded The Blood Lipids and BMI Monitoring Form.

CONTACTS AND LOCATIONS:
Locations (1):
- Gümüşhane State Hospital and Gümüşhane Kelkit State Hospital, Gümüşhane, Turkey (Türkiye)

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT05987462/Prot_SAP_ICF_000.pdf